CLINICAL TRIAL: NCT02009644
Title: A Phase II Clinical Study of the Safety and Performance of the Treovance Stent-Graft With Navitel Delivery System for Patients With Infrarenal Abdominal Aortic Aneurysms
Brief Title: Clinical Study of the Treovance Stent-Graft for Patients With Abdominal Aortic Aneurysms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0008-12
Record Dates: First submitted 2013-11-06; First posted 2013-12-12 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: Abdominal Aortic Aneurysm; AAA; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Intervention Model Description: AAA Device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treovance (Experimental): Subjects who receive the Treovance stent-graft
  Interventions: Device: Subjects who receive the Treovance stent-graft

INTERVENTIONS:
Device: Subjects who receive the Treovance stent-graft — Eligible subjects will be implanted with the Treovance Stent-Graft
  Other Names: Treovance Abdominal Stent-Graft with Navitel Delivery System

SUMMARY:
The purpose of this clinical trial is to assess and evaluate the safety and efficacy of the Treovance Stent-Graft with Navitel Delivery System in subjects with Abdominal Aortic Aneurysms (AAA).

DETAILED DESCRIPTION:
This is a phase II, multi-center, non-blinded, non-randomized study of treatment with the Treovance Stent-Graft in subjects with abdominal aortic aneurysms. The study will include 150 subjects treated with the Treovance Stent-Graft at a maximum of 30 investigational sites. Upon completion of enrollment of150 subjects, an additional 50 subjects may be treated with the Treovance Stent-Graft at the 30 investigative sites participating in the trial. These additional subjects will follow the same study schedule, and data from these patients may be used to supplement the pivotal trial data. There will be no prospective control group. Subjects diagnosed with infrarenal abdominal aortic aneurysms enrolled in the trial will be treated with the Treovance Stent-Graft with Navitel Delivery System. Pre-procedure baseline data will be gathered, as well as post-procedure assessments prior to hospital discharge and 30 days, 6 months, and 12 months post-implantation. In addition, annual follow-up visits out to 5 years will be conducted. Subjects with fracture(s) confirmed by the Core Lab within the first 5 years will be followed for an additional 5 years, for a total of 10 years post-implantation.

The primary goal of this study is to gather safety and effectiveness data on the Treovance device. A maximum of 150 endovascular subjects will be required to fulfill the U.S. Phase II requirements. The data from this study will be submitted to the FDA and used to support approval in the U.S.

There are two primary objectives, efficacy and safety of the Treovance Stent-Graft in subjects with infrarenal aortic aneurysms:

* Primary Efficacy will be evaluated by successful aneurysm treatment 12 months post-implant
* Primary Safety will be assessed by composite major adverse event (MAE) rate at 30-days

Secondary objectives involve assessment of major device-related events and major morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be between the ages of 18 and 85
2. Subject must be diagnosed with an infrarenal abdominal aortic aneurysm (AAA), with or without iliac artery involvement, by CT with contrast performed within 4 months of planned implant procedure
3. Subject must have an infrarenal AAA that i. is > 4.5 cm in diameter for males, or > 4.0 cm in diameter for females, or ii. has increased in diameter by 0.5 cm in the last 6 months
4. Subject must have i. infrarenal landing neck length of 10 mm or greater and an angle of less than 60 degrees relative to the long axis of the aneurysm (centerline at lowest renal to centerline at bifurcation) and a suprarenal neck angle of less than 45 degrees relative to the infrarenal neck axis and an outside diameter of 17 mm -32 mm, or ii. infrarenal landing neck length of 15 mm or greater and an angle of between 60 and 75 degrees relative to the long axis of the aneurysm and a suprarenal neck angle of less than 45 degrees relative to the infrarenal neck axis and an outside diameter of 16 mm-30 mm
5. Subject's infrarenal landing neck must meet the vessel size requirements specified in the instructions for use (IFU) for the corresponding devices
6. Subject must have lowest renal artery at least 9 cm from the aortic bifurcation
7. Subject must have a distal iliac landing neck with i. an inside diameter of 8 mm - 13 mm and a length of at least 10 mm, or ii. an inside diameter of >13 mm - 20 mm and a length of at least 15 mm
8. Subject's distal iliac landing neck must meet the vessel size requirements specified for the corresponding devices in the IFU
9. Subject must have a total treatment length of at least 13 cm
10. Subject must have a distal aortic diameter above the iliac bifurcation equal to or greater than 70% of the sum of the selected leg graft diameters that will pass through the same
11. Subject must be willing and able to comply with 1-month, 6-month, and 12-month follow-up visits, as well as annual visits out to 5 years
12. Subject must have adequate renal function to tolerate required follow-up contrast-enhanced CTs
13. Subject must have adequate vascular access (e.g., patent iliac or femoral arteries) for introduction of the Navitel Delivery System, which is 18F (6 mm) or 19F (6.3 mm) outer diameter based on size of device used. Alternatively, subject's anatomy is suitable for creation of an iliac conduit.
14. Subject or Legally Authorized Representative (LAR) must agree to sign Informed Consent Form

Exclusion Criteria:

1. Subject is pregnant or lactating
2. Subject has a dissection in abdominal aorta, ruptured aneurysm, or symptomatic aneurysm (as determined by treating physician)
3. Subject has a patent inferior mesenteric artery that cannot be sacrificed and an occluded or stenotic celiac and/or superior mesenteric artery
4. Implant procedure as planned does not allow for at least one patent hypogastric artery left intact, unless both are occluded on pre-op imaging
5. Subject has a lesion that cannot be crossed by a guide wire
6. Proximal neck cannot increase by more than 10% over 15mm or more than 7% over 10mm; i.e., no trapezoidal necks
7. Subject has severe untreated coronary artery disease and/or unstable angina, significant areas of myocardium at risk (based on coronary angiogram or radionuclide scans), left ventricular ejection fraction < 20%, or recent diagnosis of Congestive Heart Failure (CHF)
8. Subject has had a stroke or myocardial infarction within 6 months of the planned treatment date
9. Subject has chronic obstructive pulmonary disease requiring routine need for oxygen therapy outside the hospital setting (e.g., daily or nightly home use)
10. Subject has an active systemic infection or is suspected of having an active systemic infection (e.g.,AIDS/HIV, sepsis)
11. Subject is morbidly obese (more than 100% over the ideal body weight or as defined by institutional standards) or has other clinical conditions that severely compromise or impair x-ray visualization of the aorta
12. Subject has connective tissue disease (e.g., Marfan's syndrome)
13. Subject has a mycotic aneurysm
14. Subject has significant or circumferential calcification or mural thrombus in the proximal aortic neck
15. Subject has significant or circumferential calcification or mural thrombus in the distal iliac landing zone
16. Subject has significant or circumferential calcification or mural thrombus within the treatment length, which may adversely impact device patency
17. Subject has a blood coagulation disorder or bleeding diathesis, the treatment for which cannot be suspended pre- and post-repair
18. Subject is in acute or chronic renal failure (creatinine > 2.5 mg/dL) unless subject is stable on dialysis
19. Subject has less than two-year life expectancy as evidenced by factors prohibiting major medical intervention (e.g., presence of malignancy, severe cardiopulmonary disease, etc.)
20. Subject is participating in another research study, has received investigational study drug within 30 days of planned procedure, or has received an investigational device within one year of planned procedure
21. Subject is confronted with other medical, social or psychological issues that the investigator believes may interfere with study treatment or follow-up. These reasons must be documented. An example may include adherence to a theological or personal doctrine with aversion or opposition to blood transfusion.
22. Subject has had a prior AAA repair (endovascular or surgical)
23. Subject has an untreatable allergy or sensitivity to contrast media, nitinol/nickel, or polyester
24. Subject has undergone other major surgical or medical intervention within 45 days of the planned procedure or is planning to undergo other major surgical or medical intervention within 45 days post implantation (e.g., Coronary Artery Bypass Graft (CABG), organ transplantation, renal stenting, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-11-23 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy | 12 months
  Successful aneurysm treatment which is a composite of the following: Technical success at the conclusion of the procedure; absence of aneurysm enlargement; absence of device-related complications (e.g., fracture, conversion to open surgical repair, etc.)
Primary Safety | 30 days
  The primary safety endpoint is composite major adverse event (MAE) rate (including myocardial infarction, stroke, respiratory failure, etc.)

SECONDARY OUTCOMES:
Secondary Efficancy Endpoint -- Aneurysm-Related Mortality | Annually to 5-years; annually to 10-years (stent-fracture subjects only)
  Aneurysm-related mortality at 12 month and annually to 5 years; annually to 10 years for subjects with Core Lab-confirmed fracture(s)
Secondary Efficacy Endpoint -- Technical Success | 30 days
  Technical success at 30 days confirmed by an imaging modality (e.g. CT)
Secondary Efficacy Endpoint -- Clinical Utility Measures | Perioperative/Periprocedural
  Clinical utility measures (procedure time, time in the intensive care unit, length of hospital stay)
Secondary Efficacy Endpoint -- Secondary interventions | 30 days, 6 months, annually to 5-years; annually to 10-years (stent-fracture subjects only)
  The secondary efficacy endpoint includes the rate of additional procedures performed to correct the original implant
Secondary Efficacy Endpoint -- Device-Related Events | 30 days, 6 months, and annually to 5-years; annually to 10-years (stent-fracture subjects only)
  This endpoint includes the rate of events associated with the device.
Secondary Safety Endpoint -- Individual Rate for Events included in the composite MAE | 30 days, 6 months, annually to 5 years
  Secondary safety endpoints will include each individual rate for the adverse events included in the composite MAE at 30 days, 6 months, and annually to 5 years
Secondary Safety Endpoint -- Procedure-Related Complications | 30 days, 6 months, annually to 5 years
  Procedure-related complications at 30 days, 6 months, 12 months, and annually to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Eagleton, MD, Principal Investigator — Cleveland Clinic Foundaton
Locations (29):
- United States (29):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Danbury Hospital, Danbury, Connecticut
  - Lynn Heart and Vascular Institute, Boca Raton, Florida
  - Northside Hospital Heart & Vascular Institute, Atlanta, Georgia
  - Presence Medical Center -- Christie Clinic, Champaign, Illinois
  - University of Chicago, Chicago, Illinois
  - Affiliated Surgeons of Rockford Memorial Hospital, Rockford, Illinois
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - Tufts University Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Community Care (previously Albany Medical Center), Albany, New York
  - Buffalo General Medical Center, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester -- Strong Memorial Hospital, Rochester, New York
  - Stony Brook Medical Center, Stony Brook, New York
  - Mission Hospital, Asheville, North Carolina
  - East Carolina University / Pitt County Memorial Hospital, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - North Central Heart (Avera Heart Hospital), Sioux Falls, South Dakota
  - Sanford University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Sentara Vascular Specialists, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No